CLINICAL TRIAL: NCT00848978
Title: Health Enhancing Strength Training in Nonagenarians
Brief Title: Strength Training in Nonagenarians
Acronym: STRONG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Universidad Europea de Madrid (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jose Antonio Serra, MD PhD Head of Department(Geriatry), Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 140
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Elderly
Keywords: Functional capacity; Quality of life; Depression; Falls; Body composition; Physical activity
MeSH Terms: conditions — Depression; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental): The experimental group will participate in the aerobic and strength training program.
  Interventions: Behavioral: 8-week aerobic and strength training program
- 1 (No Intervention): The usual care group will receive general physical activity guidelines.

INTERVENTIONS:
Behavioral: 8-week aerobic and strength training program — Participants allocated in the intervention group will be enrolled in three weekly non-consecutive training sessions for 8 weeks. Each session will last for about 45-50 min. The exercise program will consist of muscular strength and aerobic exercises. Each session will start and end with a low intensity ~5-7 min warm-up and cool-down period respectively, consisting mainly of stretching exercises involving all major muscle groups.
  Arms: 2

SUMMARY:
The Health Enhancing Strength Training in Nonagenarians (STRONG) is a randomised control trial to assess the effectiveness of an aerobic and strength training program for improving functional capacity and quality of life in nonagenarians. Sixty (51 women) nonagenarians (age range: 90-102 years) who live in a geriatric nursing home will be randomly assigned to either a usual care (control) group (n=30) or an intervention (training) group (n=30). Participants allocated in the usual care group will receive general physical activity guidelines and participants allocated in the intervention group will also enroll in three weekly non-consecutive individualized training sessions (~45-50 min each) during 8 weeks. The exercise program will consist of muscular strength [with a special focus on leg press at 30% (start of the program) to 70% 1 repetition maximum (end)] and aerobic exercises (cycle-ergometry during 3-5 to 15 minutes at 12-14 points in the rate of perceived exertion scale). Results from STRONG will help to better understand the potential of regular physical activity for improving the well-being of the oldest population groups.

ELIGIBILITY:
Inclusion Criteria:

* Age: 90 years or over.
* Planning to stay in the same nursing home during the study.
* Able to ambulate, with or without assistance.
* Able to communicate.
* Informed consent: Must be capable and willing to provide consent.

Exclusion Criteria:

* Acute or terminal illness.
* Myocardial infarction in the past 3 months.
* Not capable to ambulate.
* Unstable cardiovascular disease or other medical condition.
* Upper or lower extremity fracture in the past 3 months.
* Severe dementia.
* Unwillingness to either complete the study requirements or to be randomised into control or training group.
* Presence of neuromuscular disease or drugs affecting neuromuscular function.

Ages: 90 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Functional capacity and quality of life | August 2009

SECONDARY OUTCOMES:
Depressive symptoms, falls and body composition | August 2009

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

REFERENCES:
- [Derived] Serra Rexach JA, Ruiz JR, Bustamante-Ara N, Villaran MH, Gil PG, Sanz Ibanez MJ, Sanz NB, Santamaria VO, Sanz NG, Prada AB, Gallardo C, Romo GR, Lucia A. Health enhancing strength training in nonagenarians (STRONG): rationale, design and methods. BMC Public Health. 2009 May 26;9:152. doi: 10.1186/1471-2458-9-152. PMID 19470176